CLINICAL TRIAL: NCT06044766
Title: A Clinical Study to Verify the Reliability of Root Form Classification of Impacted Lower Third Molars
Brief Title: Verification of the Root Form Classification of Impacted Lower Third Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Nedal Abu-Mostafa, Assistant Professor in Oral and Maxillofacial Surgery, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REU2
Record Dates: First submitted 2023-05-11; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Impacted Lower Third Molars Roots
Keywords: impacted lower third olars; Roots morphology; Root forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical exatrction of impacted lower third molars (Other): Clinical intervention: Surgical exatrction of impacted lower third molar to examine and classify the roots, then to compare it with radiographic classification
  Interventions: Procedure: Surgical exatrction of impacted lower third molars

INTERVENTIONS:
Procedure: Surgical exatrction of impacted lower third molars — Surgical exatrction of impacted lower third molars to verify the form of the root

SUMMARY:
A clinical study will be conducted to verify the reliability of the root form classification of impacted lower third molars that was put by Abu-Mostafa N (2023) The root forms of partially or fully impacted lower third molars will be classified pre-operatively based on panoramic radiograph, then clinically after extraction, and the identified root classifications will be compared.

DETAILED DESCRIPTION:
According to Abu-Mostafa N, the roots of impacted lower third molars are classified into two types: Fused roots and separated roots. Both have different forms:

Fused roots forms: Straight, Curved distal, Curved mesial, and S-shaped.

Separated roots forms: Straight, Both roots are curved distal, Both roots are curved mesial, Joined roots, One root is straight and one is curved, and More than two roots.

A panoramic radiograph will be taken before extraction, then the roots will be classified by two Oral biologist and Oral and Maxillofacial Surgeon individually. After surgical extraction of the third molar, the roots will be examined clinically and classified according to the same classification.

The two pre-extraction radiographic classifications will be compared together, and then they will be compared with the clinical classification to check if there is a discrepancy.

The surgical extraction procedure:

Local anesthesia will be achieved by inferior alveolar nerve block and buccal infiltration using Lidocaine 2% with Epinephrine 1:100,000. A flap with a distobuccal releasing incision will be done. The bone reduction will be performed by a low-speed surgical handpiece under irrigation with normal saline. Root separation is done of required for the third molars with separated root forms. The tooth will be luxated by straight elevators and then extracted.

The evaluation results will be categorized to:

* Agreement: The two pre-extraction radiographic evaluations and the clinical evaluations are similar
* Discrepancy 1: One pre-extraction radiographic evaluation and the clinical evaluations are similar, but the other radiographic evaluation differs.
* Discrepancy 2: the two pre-extraction radiographic evaluations are similar, but the clinical evaluation differs.
* Disagreement: The three evaluations are different

The results will be analyzed regarding frequencies and association of each category with root forms

ELIGIBILITY:
Inclusion Criteria:

Patients with impacted lower third molars who visit Riyadh Elm University" hospital and have lower third molars which are diagnosed clinically and radiographically as partially or fully impacted. The roots of these third molars have to be fully formed.

Exclusion Criteria:

incomplete apex formation and root resorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Frequency of discrepancies and agreements on the classified root forms | Before surgical exatration
  To report the radiographic classifications of root forms by two examiners
Frequency of discrepancies and agreements on the classified root forms | Immidiately after extraction
  To report the clinical classifications of root forms

SECONDARY OUTCOMES:
The frequency of root types | Immediately after extraction
  The frequency of fused roots and separated roots
The frquency of fused root forms | Immediately after extraction
  The frequency of the four fused roots forms
The frequency of separated root forms | Immediately after extraction
  The frequency of the six separated root forms

IPD SHARING:
Plan to Share IPD: No
After publication